CLINICAL TRIAL: NCT00520039
Title: Effect of Osteopathic Manipulative Medicine (OMM) on the Duration of Middle Ear Effusion in Children Following Diagnosis of Acute Otitis Media, as Measured by Tympanograms and Acoustic Reflectometry
Brief Title: Osteopathic Otitis Media Research Study
Acronym: OOMRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia School of Osteopathic Medicine (Other)
Collaborators: University of New England (Other); American Academy of Osteopathy (Other); Osteopathic Research Center (Unknown)
Responsible Party: Principal Investigator, Karen M. Steele, D.O., FAAO, Professor Emerita, West Virginia School of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KS5172007
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2017-08

CONDITIONS: Otitis Media With Effusion
Keywords: Otitis Media; Effusion; OMM; OMT; Resolution
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care Plus OMM (Experimental): Subjects will receive active intervention with osteopathic manipulative medicine (OMM) using a prescribed standardized treatment protocol which is age appropriate. Subjects will also receive standard care for otitis media from their referring physician.
  Interventions: Procedure: osteopathic manipulative medicine (OMM)
- Standard Care Only (No Intervention): Subjects will receive standard care only for otitis media from their regular referring physician

INTERVENTIONS:
Procedure: osteopathic manipulative medicine (OMM) — At each of the first three study visits, all subjects in the osteopathic manipulative medicine (OMM) group will receive OMM using the prescribed protocol.
  Arms: Standard Care Plus OMM

SUMMARY:
The purpose of this study is to determine if the application of osteopathic manipulative medicine speeds the rate of resolution of middle ear effusion (fluid) in children following an episode of acute otitis media.

DETAILED DESCRIPTION:
Acute otitis media is a significant world wide problem commonly affecting children between 6 and 18 months, and is the most frequent reason for childhood illness visits to a physician in the US. By three years of age, 50-70% of children will have had one episode, while one-third will have had more than three. Persistence of middle ear effusion following an episode of acute otitis media is thought to predispose the child to recurrent infection. The standard care for recurrent acute otitis media includes long term antibiotic prophylaxis and surgery. The risks of standard care are recognized, and alternative means of treating acute disease and preventing recurrent otitis media are needed.

For over a century, osteopathic physicians have reported favorable clinical outcomes in children treated with osteopathic manipulative medicine (OMM) in addition to standard medical care. To determine if a standardized OMM protocol will reduce the duration of middle ear effusion (MEE) after onset of acute otitis media, we outline a prospective, randomized, blinded, multi-center efficacy study of children ages six months to two years with a single episode of acute otitis media. Subjects will be randomized into one of two treatment groups: standard care plus OMM and standard care only. Subjects will be followed for one month to determine rate of resolution of middle ear effusion following onset of the acute otitis media. Statistical analysis will determine any differences between subjects in the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months up to second birthday
* Documented presence of acute otitis media following the 2004 AAP/AAFP Guidelines within 3 days of entry into the study

Exclusion Criteria:

* Chromosomal abnormalities
* Major congenital malformations of the head and neck, including torticollis
* Immunologic abnormalities or deficiencies
* Any prior ear-nose-throat surgery performed as a treatment for otitis media
* Any tube placement surgery scheduled during the four weeks of the study.
* Normal tympanograms at entry into study

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Steele, D.O., Principal Investigator — West Virginia School of Osteopathic Medicine
Locations (2):
- United States (2):
  - University of New England College of Osteopathic Medicine, Biddeford, Maine
  - West Virginia School of Osteopathic Medicine, Lewisburg, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steele KM, Carreiro JE, Viola JH, Conte JA, Ridpath LC. Effect of osteopathic manipulative treatment on middle ear effusion following acute otitis media in young children: a pilot study. J Am Osteopath Assoc. 2014 Jun;114(6):436-47. doi: 10.7556/jaoa.2014.094. PMID 24917631
- [Derived] Steele KM, Viola J, Burns E, Carreiro JE. Brief report of a clinical trial on the duration of middle ear effusion in young children using a standardized osteopathic manipulative medicine protocol. J Am Osteopath Assoc. 2010 May;110(5):278-84. PMID 20538749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: September 2007 through May 2009 Site: medical clinics of 2 colleges of osteopathic medicine Location: mid-Atlantic and Northeast areas of the United States
Pre-assignment Details: 52 subjects were enrolled and randomized into the two study groups. 5 subjects in the SCO group and 7 subjects in the SC+OMM group were excluded from the study due to having a normal tympanogram on the first study visit.
Groups:
- Standard Care Plus OMM (SC+OMM): Subjects will receive active intervention with osteopathic manipulative medicine (OMM) using a prescribed standardized treatment protocol which is age appropriate. Subjects will also receive standard care for otitis media from their referring physician.
  osteopathic manipulative medicine (OMM): At each of the first three study visits, all subjects in the osteopathic manipulative medicine (OMM) group will receive OMM using the prescribed protocol.
- Standard Care Only (SCO): Subjects will receive standard care only for otitis media from their regular referring physician
Period: Overall Study
Arm/Group | Standard Care Plus OMM (SC+OMM) | Standard Care Only (SCO)
Started | 28 | 24
Completed | 21 | 19
Not Completed | 7 | 5
Not completed — Exclusion criteria met at first visit | 7 | 5

BASELINE CHARACTERISTICS:
Population: 52 participants were enrolled and 12 excluded due to normal tympanograms at first study visit, leaving 19 subjects in the SCO and 21 subjects in the SC+OMM group.
Groups:
- Standard Care Plus OMM: Subjects will receive active intervention with osteopathic manipulative medicine (OMM) using a prescribed standardized treatment protocol which is age appropriate, at each of the first 3 study visits. Subjects will also receive standard care for otitis media from their referring physician.
- Total: Total of all reporting groups
Arm/Group | Standard Care Plus OMM | Standard Care Only | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 24 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 16 | 13 | 29
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Middle Ear Effusion Over Four Weeks Following an Episode of Acute Otitis Media
Description: For this study, the tympanogram was chosen to measure middle ear effusion. Three tympanogram readings from each ear included in the study were taken at the beginning of each of 5 Study Visits. For the intervention group, a second set of 3 tympanograms was taken immediately after the OMM on Visits 1, 2 and 3. All tympanograms were sent to a blinded audiologist, who chose the most healthy of the 3 tympanogram readings for interpretation, rating it according to standard protocols. "A" and "C1" readings were considered "normal" and "B" and "C2" readings were considered "abnormal". The extent to which the tympanogram readings of each ear included in the study changed from baseline over 4 weeks was computed by crosstabulating the intervention group by the normal/abnormal changes in tympanograms.
Time Frame: 1 month
Population: 4 ears, from 2 subjects, were removed from the SC+OMM group final analysis due to no interpretable readings obtained during the study.
Measure: Number; unit: Ears
Units Other Than Participants: Ears
Arm/Group | Standard Care Plus OMM (SC+OMM) | Standard Care Only (SCO)
Number analyzed (Participants) | 19 | 19
Number analyzed (Ears) | 38 | 38
Ears
  Improvement in MEE at 2 weeks | 26 | 16
  No Improvement in MEE at 2 weeks | 12 | 22
Statistical Analysis 1: Comparison: Standard Care Plus OMM (SC+OMM) vs Standard Care Only (SCO); Test of the null hypothesis that there is no improvement in MEE at Visit 3 using tympanogram; Test type: Superiority or Other; p = 0.02, Chi-squared; df = 1; Odds Ratio, log = 1.09, 95% CI 2-sided [0.15 to 2.03], Standard Error of Mean 0.94 — The denominator of the Odds ratio represents the odds of improvement for the Standard Care Only (SCO) group

2. Secondary Outcome: Change in Middle Ear Effusion Immediately After OMM at Study Visit 2
Description: For this study, the tympanogram was chosen to measure middle ear effusion. For the SC+OMT Group during study visit 2, three tympanogram readings from each ear included in the study were taken prior to, and immediately after the intervention. The tympanograms were sent to the blinded audiologist, who chose the most healthy of the 3 tympanogram readings for interpretation, rating it according to standard protocols. "A" and "C1" readings were considered "normal" and "B" and "C2" readings were considered "abnormal". The extent to which the tympanogram readings of each ear included in the study changed between "normal" and "abnormal" from before and after the OMM was computed.
Time Frame: Before and immediately after OMM at study visit 2
Measure: Number; unit: ears
Units Other Than Participants: ears
Groups:
- Before OMM: Result of tympanogram reading before OMM.
  Subjects will receive active intervention with osteopathic manipulative medicine (OMM) using a prescribed standardized treatment protocol which is age appropriate. Subjects will also receive standard care for otitis media from their referring physician.
- After OMM: Result of tympanogram reading after OMM.
  Subjects will receive active intervention with osteopathic manipulative medicine (OMM) using a prescribed standardized treatment protocol which is age appropriate. Subjects will also receive standard care for otitis media from their referring physician.
Arm/Group | Before OMM | After OMM
Number analyzed (Participants) | 19 | 19
Number analyzed (ears) | 31 | 29
ears
  Resolution of MEE after OMM at Visit 2 | 5 | 6
  No Resolution of MEE at end of OMM at visit 2 | 26 | 23
Statistical Analysis 1: Comparison: Before OMM vs After OMM; Test type: Superiority or Other; p = 0.32, Chi-squared; df = 1; Odds Ratio, log = 0.31, 95% CI 2-sided [-1.00 to 1.62], Standard Error of Mean 1.31 — The odds of Resolution of MEE before OMT is represented in the denominator of the odds ratio

3. Secondary Outcome: Change in Middle Ear Effusion Immediately After OMM at Study Visit 3
Description: For this study, the tympanogram was chosen to measure middle ear effusion. For the SC+OMT Group during study visit 3, three tympanogram readings from each ear included in the study were taken prior to, and immediately after the intervention. The tympanograms were sent to the blinded audiologist, who chose the most healthy of the 3 tympanogram readings for interpretation, rating it according to standard protocols. "A" and "C1" readings were considered "normal" and "B" and "C2" readings were considered "abnormal". The extent to which the tympanogram readings of each ear included in the study changed between "normal" and "abnormal" from before and after the OMM was computed.
Time Frame: Before and immediately after OMM at study visit 3
Measure: Number; unit: ears
Units Other Than Participants: ears
Arm/Group | Before OMM | After OMM
Number analyzed (Participants) | 19 | 19
Number analyzed (ears) | 31 | 29
ears
  Resolution of MEE at Visit 3 | 12 | 13
  No Resolution of MEE after OMM at Visit 3 | 19 | 25
Statistical Analysis 1: Comparison: Before OMM vs After OMM; Test type: Superiority or Other; p = .31, Chi-squared; df = 1; Odds Ratio, log = 0.25, 95% CI 2-sided [-0.78 to 1.28], Standard Error of Mean 1.03

ADVERSE EVENTS:
Time Frame: 1month
Description: Completed at the start of each study visit by the Research Assistant, and during the intervention by the OMM treatment provider
Groups:
- Standard Care Plus OMM: Subjects will receive active intervention with osteopathic manipulative medicine (OMM) using a prescribed standardized treatment protocol which is age appropriate. Subjects will also receive standard care for otitis media from their referring physician.
  osteopathic manipulative medicine (OMM): At each of the first three study visits, all subjects in the osteopathic manipulative medicine (OMM) group will receive OMM using the prescribed protocol.
  There were no Serious Adverse Events reported.
- Standard Care Only: Subjects will receive standard care only for otitis media from their regular referring physician.
  There were no Serious Adverse Events reported.
Arm/Group | Standard Care Plus OMM | Standard Care Only
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/24
Other Adverse Events (participants affected / at risk) | 0/28 | 0/24

LIMITATIONS AND CAVEATS:
One site closed after year 1 due to lower than expected subject recruitment. Lower than expected recruitment overall.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No